CLINICAL TRIAL: NCT07367347
Title: The Effect of Increased BMI on Efficacy of Labor Analgesia: A Retrospective Cohort Study
Brief Title: Effect of Increased BMI on Efficacy of Labor Analgesia
Status: Completed | Type: Observational
Sponsor: Mariah Arif (Other Government)
Responsible Party: Sponsor-Investigator, Mariah Arif, Resident Physician, Hamad General Hospital
Organization: Hamad General Hospital (Other Government)
Other Study IDs: MRC-01-24-875
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Neuraxial Analgesia; Labor Analgesia
Keywords: labor analgesia; neuraxial analgesia; obesity; parturient
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Class III obese parturient: Class III obese parturient receiving neuraxial analgesia
  Interventions: Procedure: Neuraxial analgesia

INTERVENTIONS:
Procedure: Neuraxial analgesia — Combined spinal-epidural analgesia
Procedure: Neuraxial Analgesia — Epidural analgesia
Procedure: Neuraxial Analgesia — Dural puncture epidural analgesia

SUMMARY:
This study seeks to identify the most effective neuraxial technique for labor analgesia in Class III parturient

DETAILED DESCRIPTION:
This retrospective cohort study collected data on eligible participants from the electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* BMI ≥ 40 kg/m²
* Gestational age ≥ 28 weeks

Exclusion Criteria:

* Age < 18 years
* BMI < 40 kg/m²
* History of venous thromboembolism or arterial disease (e.g., DVT, PE, angina, MI, or stroke)
* Severe active lung, cardiovascular, renal, or liver disorders; autoimmune disease; or hemoglobinopathies
* Hereditary or acquired thrombophilia (e.g., Factor V Leiden mutation or antithrombin deficiency)
* In utero fetal demise (IUFD)
* Failed operative vaginal delivery
* Cesarean for the second twin or multiple pregnancies (triplets or higher)
* IVF pregnancy
* Intraoperative bleeding>1500mL
* Emergency cesarean section (Category I)
* Presence of large uterine fibroid ≥10 cm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Class III obese parturient receiving neuraxial analgesia (CSE, epidural or DPE) in labor rooms of Women's Wellness and Research Center between 1 January 2015 to 1 December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Success rate of labor analgesia | onset of neuraxial analgesia to completion of labor
  The success rate of each technique will be determined by:
  Number of patients requiring a physician top-up bolus Block symmetry First-attempt success rate

SECONDARY OUTCOMES:
Maternal adverse events | onset of neuraxial analgesia to completion of labor
  Incidence of maternal hypotension, maternal bradycardia, high block (above T1), higher than T4 block, need of vasopressors, mortality, post-Dural puncture headache
Fetal adverse events | at 1 and 5 minutes after birth
  APGAR SCORE

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Saracoglu, Principal Investigator — University of Florida, UF Health, Jacksonville, FL 32209, USA
Locations (1):
- Women's Wellness and Research Center, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No